CLINICAL TRIAL: NCT02825927
Title: Swallowing Function, Oral Health, and Food Intake in Old Age
Acronym: SOFIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Örebro County (Other); Karlstad University (Other); Region Gävleborg (Other); Dalarna University (Other); Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/100/3
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2016-06

CONDITIONS: Dysphagia; Deglutition Disorders; Swallowing Disorders; Quality of Life
Keywords: Dysphagia; Oral screen; Intervention; Oral Health; Food Intake; Quality of life; Elderly; Short-term care facilities
MeSH Terms: conditions — Deglutition Disorders | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intensive training with oral screen for 5 weeks.
  Interventions: Other: Oral screen
- Control group (No Intervention): The control group is not offered any intervention.

INTERVENTIONS:
Other: Oral screen — The oral screen is used for 30 seconds, three times a day, before meals and implies new possibilities for training of the orofacial muscles.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine whether a specific rehabilitation program with oral screen used in an elderly population with dysphagia can improve elderly's swallowing capacity.

DETAILED DESCRIPTION:
The present study aims to investigate the effects on swallowing function of a specific rehabilitation program with oral screen in the elderly population included. The present study is a part of an on-going cross-sectional, descriptive project called SOFIA where approximately 400 elderly individuals, admitted to short-term care (from the five regions/county Dalarna, Gävleborg, Örebro, Värmland and Västerbotten in Sweden), will be included. The purpose of the overall project is to gain a broader understanding of aspects of dysphagia, eating, oral health, and quality of life and care among elderly people in short-term care facilities.

In the present study, 35 elderly individuals identified with dysphagia in the overall project (swallowing capacity <10ml/sec) and without known dementia will be offered to participate and to undergo oral screen training for 5 weeks. The participants' status regarding swallowing, eating, quality of life and oral health will be assessed before and immediately after the intervention and 6-months post-intervention. A control group (35 people in short-term accommodation included in the overall project, identified with dysphagia but not offered the intervention) will undergo the same assessments (at start, after 5 weeks, and 6-month post-intervention) as the intervention group regarding swallowing, eating, quality of life and oral health status.

Cluster randomisation of short-term accommodation facilities will be made for those patients participating from the five regions/county to either intervention group or control group. Participants will be recruited consecutively to either the intervention- or the control group, depending on which short-term care facility they are staying at.

The investigators hypothesize that oral screen rehabilitation for elderly individuals with dysphagia and with different diagnoses treated in short-term care results in improved swallowing capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Admitted to short-term care facility ≥ 3 days
* Included in the overall project SOFIA and with a swallowing capacity <10ml/sec

Exclusion Criteria:

* Incapable of making decisions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Swallowing function | Baseline, 5 weeks and 6 months post-intervention
  Change in swallowing function measured by the Swallowing Capacity Test (SCT) combined with a teaspoon test. Comparisons between intervention-and control group will be made.

SECONDARY OUTCOMES:
Quality of life related to swallowing | Baseline, 5 weeks and 6 months post-intervention
  Change in quality of life related to swallowing measured by the Swallowing Quality of Life Questionnaire (SWAL-QOL). Comparisons between intervention-and control group will be made.
Oral Health | Baseline, 5 weeks and 6 months post-intervention
  Change in oral health status measured by the Revised Oral Assessment Guide (ROAG). Comparisons between intervention-and control group will be made.
Food Intake | Baseline, 5 weeks and 6 months post-intervention
  Change in nutritional status measured by the Minimal Eating Observation and Nutrition Test Version II ( MEONF-II). Comparisons between intervention-and control group will be made.
Activity of daily living | Baseline, 5 weeks and 6 months post-intervention
  Change in status regarding activity of daily living measured by the Katz Index of Independence in Activities of Daily Living (Katz ADL-index). Comparisons between intervention-and control group will be made.
Quality of life related to oral health | Baseline, 5 weeks and 6 months post-intervention
  Change in quality of life related to oral health measured by the Oral Health Impact Profile (OHIP-14). Comparisons between intervention-and control group will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Carlsson, PhD, Nurse, Principal Investigator — Region Örebro
Locations (1):
- Region Örebro län, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagglund P, Hagg M, Wester P, Levring Jaghagen E. Effects of oral neuromuscular training on swallowing dysfunction among older people in intermediate care-a cluster randomised, controlled trial. Age Ageing. 2019 Jul 1;48(4):533-540. doi: 10.1093/ageing/afz042. PMID 31062842
- [Derived] Hagglund P, Falt A, Hagg M, Wester P, Levring Jaghagen E. Swallowing dysfunction as risk factor for undernutrition in older people admitted to Swedish short-term care: a cross-sectional study. Aging Clin Exp Res. 2019 Jan;31(1):85-94. doi: 10.1007/s40520-018-0944-7. Epub 2018 Apr 16. PMID 29663160
- [Derived] Hagglund P, Olai L, Stahlnacke K, Persenius M, Hagg M, Andersson M, Koistinen S, Carlsson E. Study protocol for the SOFIA project: Swallowing function, Oral health, and Food Intake in old Age: a descriptive study with a cluster randomized trial. BMC Geriatr. 2017 Mar 23;17(1):78. doi: 10.1186/s12877-017-0466-8. PMID 28335729